CLINICAL TRIAL: NCT06311045
Title: Basis of Sex-specific Therapeutic Responses to Obstructive Sleep Apnea (OSA): a Trial of N-acetylcysteine (NAC) in Obstructive Sleep Apnea (OSA)
Brief Title: Obstructive Sleep Apnea (OSA) and Sex-Specific Responses to N-acetylcysteine (NAC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 23-01469
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Acetylcysteine; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAC (Experimental): Following run-in PAP therapy per standard clinical care for 12 weeks, participants randomized to the NAC arm will also receive the supplement N-acetylcysteine (NAC) for four weeks while remaining on PAP therapy.
  Interventions: Dietary Supplement: N-acetylcysteine (NAC); Procedure: Positive Airway Pressure (PAP) Therapy
- Placebo (Experimental): Following run-in PAP therapy per standard clinical care for 12 weeks, participants randomized to the placebo arm will also receive placebo for four weeks while remaining on PAP therapy.
  Interventions: Dietary Supplement: Placebo; Procedure: Positive Airway Pressure (PAP) Therapy

INTERVENTIONS:
Dietary Supplement: N-acetylcysteine (NAC) — Participants will take two NAC 600mg capsules daily for four weeks.
  Arms: NAC
Dietary Supplement: Placebo — Participants will take two placebo 600mg capsules daily for four weeks.
  Arms: Placebo
Procedure: Positive Airway Pressure (PAP) Therapy — All participants will receive PAP therapy per standard of care for OSA.

SUMMARY:
This is a randomized controlled trial (RCT) of 4 weeks of study supplement N-acetylcysteine (NAC) versus placebo in persons with significant obstructive sleep apnea (OSA) who are receiving positive airway pressure therapy (PAP), the standard of care therapy. The purpose of the study is to determine if NAC is associated with sex-specific changes in overnight oxidative stress, inflammation, as well as endothelial dysfunction in persons with OSA.

ELIGIBILITY:
Inclusion Criteria:

* Apnea-hypopnea index ≥15 events/hr on portable sleep monitoring
* HbA1c <6.5%

Exclusion Criteria:

* Body mass index (BMI) ≥40 kg/m2;
* Diagnosis of diabetes mellitus, defined as the use of any diabetes medication (including glucagon like peptide [GLP]-1 agonists) currently or in the previous three months or HbA1c ≥6.5%;
* Shift work (i.e., working hours that routinely cause sleep initiation after 1:00 a.m.);
* Another major sleep disorder (i.e., circadian rhythm disorder, any history of narcolepsy, concurrently diagnosed or medication-treated restless legs syndrome, concurrently diagnosed or medication-treated chronic insomnia with the exception of antidepressant therapy);
* Regular use (more than twice/week) of an opioid/narcotic, benzodiazepine, or prescription sleep medication other than antidepressants currently or within the last month;
* The use of N-acetylcysteine in any form (oral, intravenous, inhaled) in the last seven days
* The use of other over-the-counter antioxidant therapies including vitamin C or vitamin E in the preceding 10 days
* History of reduced ejection fraction heart failure, or chronic cardiac arrhythmia requiring medication or treatment;
* Unstable or uncontrolled medical or psychiatric comorbidity requiring hospitalization or change in medication during the previous three months;
* Use of biologics or immune modulators in the last year;
* Use of systemic steroids during the previous three months;
* Current tobacco smoking;
* Inability to sign informed consent;
* Currently use of positive airway pressure therapy or another OSA treatment (e.g., hypoglossal nerve stimulator, oral device);
* Recent history of alcoholism or drug abuse (within the last three months)
* Neurological condition that requires ongoing pharmacological therapy (e.g., Parkinson's disease, Alzheimer's dementia, multiple sclerosis, other degenerative neurological disease).
* Pregnancy

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Overnight Levels of Glutathione (GSH) | Baseline, Final Study Visit (4 Weeks post Initiation of Study Therapy; up to Month 6)
  GSH measured using participant blood samples.
Mean Change in Pre- to Post-Sleep GSH Levels | Baseline
  GSH measured using participant blood samples.
Mean Change in Pre- to Post-Sleep GSH Levels | Final Study Visit (4 Weeks post Initiation of Study Therapy; up to Month 6)
  GSH measured using participant blood samples.

SECONDARY OUTCOMES:
Ratio of GSH to oxidized GSH (GSSG) (GSH:GSSG) | Baseline
  GSH:GSSG measured using participant blood samples.
Ratio of GSH to oxidized GSH (GSSG) (GSH:GSSG) | Final Study Visit (4 Weeks post Initiation of Study Therapy; up to Month 6)
  GSH:GSSG measured using participant blood samples.
8-Isoprostane Level | Baseline
  8-isoprostane levels measured using participant blood samples.
8-Isoprostane Level | Final Study Visit (4 Weeks post Initiation of Study Therapy; up to Month 6)
  8-isoprostane levels measured using participant blood samples.
Plasma Nitrate Level | Baseline
  Plasma nitrate levels measured using participant blood samples.
Plasma Nitrate Level | Final Study Visit (4 Weeks post Initiation of Study Therapy; up to Month 6)
  Plasma nitrate levels measured using participant blood samples.
Plasma Nitrite Level | Baseline
  Plasma nitrite levels measured using participant blood samples.
Plasma Nitrite Level | Final Study Visit (4 Weeks post Initiation of Study Therapy; up to Month 6)
  Plasma nitrite levels measured using participant blood samples.
Organic Nitrite Level | Baseline
  Organic nitrite levels measured using participant blood samples.
Organic Nitrite Level | Final Study Visit (4 Weeks post Initiation of Study Therapy; up to Month 6)
  Organic nitrite levels measured using participant blood samples.
Interleukin 6 (IL-6) Level | Baseline
  IL-6 levels measured using participant blood samples.
Interleukin 6 (IL-6) Level | Final Study Visit (4 Weeks post Initiation of Study Therapy; up to Month 6)
  IL-6 levels measured using participant blood samples.
Tumor Necrosis Factor-alpha (TNFα) Receptor-1 (TNFα-R1) Level | Baseline
  TNFα-R1 levels measured using participant blood samples.
Tumor Necrosis Factor-alpha (TNFα) Receptor-1 (TNFα-R1) Level | Final Study Visit (4 Weeks post Initiation of Study Therapy; up to Month 6)
  TNFα-R1 levels measured using participant blood samples.
Tumor Necrosis Factor-alpha (TNFα) Receptor-2 (TNFα-R2) Level | Baseline
  TNFα-R2 levels measured using participant blood samples.
Tumor Necrosis Factor-alpha (TNFα) Receptor-2 (TNFα-R2) Level | Final Study Visit (4 Weeks post Initiation of Study Therapy; up to Month 6)
  TNFα-R2 levels measured using participant blood samples.
Reactive Hyperemia Index (RHI) Score | Baseline
  RHI is a measure of endothelial-dependent vasodilation and is assessed using a noninvasive vascular tone measure (EndoPAT®). RHI reflects endothelial health, with lower scores signifying more dysfunction. RHI less than 1.67 is considered a sign of endothelial dysfunction and RHI equal to or greater than 1.67 is considered normal function.
Reactive Hyperemia Index (RHI) Score | Final Study Visit (4 Weeks post Initiation of Study Therapy; up to Month 6)
  RHI is a measure of endothelial-dependent vasodilation and is assessed using a noninvasive vascular tone measure (EndoPAT®). RHI reflects endothelial health, with lower scores signifying more dysfunction. RHI less than 1.67 is considered a sign of endothelial dysfunction and RHI equal to or greater than 1.67 is considered normal function.
Epworth Sleepiness Scale (ESS) Score | Baseline
  ESS is an 8-item questionnaire assessing usual likelihood of falling asleep during each of eight common activities. Each item is rated on a Likert scale from 0-3. The total score is the sum of responses and ranges from 0-24; higher scores indicate greater subjective daytime sleepiness.
Epworth Sleepiness Scale (ESS) Score | Final Study Visit (4 Weeks post Initiation of Study Therapy; up to Month 6)
  ESS is an 8-item questionnaire assessing usual likelihood of falling asleep during each of eight common activities. Each item is rated on a Likert scale from 0-3. The total score is the sum of responses and ranges from 0-24; higher scores indicate greater subjective daytime sleepiness.
Insomnia Severity Index (ISI) Score | Baseline
  ISI is a 7-item questionnaire assessing the nature, severity, and impact of insomnia. Each item is rated on a 5-point Likert scale from 0-4. The total score is the sum of responses and ranges from 0-28. Scores are interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); or severe insomnia (21-28).
Insomnia Severity Index (ISI) Score | Final Study Visit (4 Weeks post Initiation of Study Therapy; up to Month 6)
  ISI is a 7-item questionnaire assessing the nature, severity, and impact of insomnia. Each item is rated on a 5-point Likert scale from 0-4. The total score is the sum of responses and ranges from 0-28. Scores are interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); or severe insomnia (22-28).
Fatigue Severity Scale (FSS) Score | Baseline
  FSS is a 9-item measure of fatigue severity from a variety of medical and neurological disorders. Each item is rated on a Likert scale from 1-7. The total score is the sum of responses and ranges from 9-63, with higher scores indicating greater fatigue.
Fatigue Severity Scale (FSS) Score | Final Study Visit (4 Weeks post Initiation of Study Therapy; up to Month 6)
  FSS is a 9-item measure of fatigue severity from a variety of medical and neurological disorders. Each item is rated on a Likert scale from 1-7. The total score is the sum of responses and ranges from 9-63, with higher scores indicating greater fatigue.
Pittsburgh Sleep Quality Index (PSQI) Score | Baseline
  PSQI is a 19-item questionnaire that is routinely used in both clinical and research settings to assess sleep quality over the preceding one month. The total score ranges from 0-21, with higher scores reflecting worse sleep quality.
Pittsburgh Sleep Quality Index (PSQI) Score | Final Study Visit (4 Weeks post Initiation of Study Therapy; up to Month 6)
  PSQI is a 19-item questionnaire that is routinely used in both clinical and research settings to assess sleep quality over the preceding one month. The total score ranges from 0-21, with higher scores reflecting worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Nisha Aurora, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Rashmi.aurora@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research. Requests should be directed to Rashmi.aurora@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request.